CLINICAL TRIAL: NCT06542627
Title: Continuous Glucose Monitoring for Glucose and Weight Management in Prediabetes and Non-severe Type 2 Diabetes
Brief Title: Continuous Glucose Monitoring for Glucose and Weight Management in Prediabetes and Non-severe Type 2 Diabetes: A Prospective Community-based (Workplace) Cohort Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Collaborators: Samsung Electronics (Industry)
Responsible Party: Principal Investigator, Cheol-Young Park, Professor, MD. PhD, Kangbuk Samsung Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KBSMC 2023-05-010
Record Dates: First submitted 2024-08-01; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: PreDiabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CGM arm (Experimental): Glycemic control was monitored using CGM data for two weeks, followed by individualized dietary education.
  Interventions: Device: Freestyle Libre

INTERVENTIONS:
Device: Freestyle Libre — Glycemic control was monitored using CGM data for two weeks, followed by individualized dietary education.

SUMMARY:
This study aimed to evaluate the effectiveness of use of Continuous Glucose Monitoring (CGM), combined with personalized dietary education and use of smartphone applications in improving glucose control and weight management.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over the age of 19
* Patients with type 2 diabetes

  * Fasting blood glucose ≥ 126 mg/dL or
  * HbA1c ≥ 6.5% or
  * Type 2 diabetes by clinical history and treated with antidiabetic medications or lifestyle Modifications
* Patients with prediabetes

  * Fasting blood glucose 100-125 mg/dL
  * HbA1c 5.7-6.4%
* Willing to participate in the study

Exclusion Criteria:

* Subjects less than 19 years old
* Patients with type 1 diabetes
* Pregnant at the time of screening or planning to become pregnant during the study
* Severe chronic diseases such as cancer, stroke, proliferative retinopathy, myocardial infarction, chronic renal disease, or amputation of a diabetic foot
* Diagnosed with or treated for myocardial infarction, stroke, end-stage renal disease, liver failure, or chronic lung disease within the past year
* Severe liver disease (e.g., cancer, liver cirrhosis, hepatitis B, hepatitis C)
* Diseases of the biliary tract, thyroid disorders, autoimmune disorders, or acute infections
* Planning to be admitted to a hospital within 2 months
* Unable to participate in the mobile intervention study as determined by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 8weeks after intervention
  HbA1c assessed by blood test after 2-week use of CGM and dietary education

SECONDARY OUTCOMES:
Fasting blood glucose | 8weeks after intervention
  Fasting blood glucose, assessed by blood test after 2-week use of CGM and dietary education
Lipid profiles | 8weeks after intervention
  Lipid profiles (total cholesterol, LDL-cholesterol, HDL-cholesterol, triglyceride), assessed by blood test after 2-week use of CGM and dietary education
Body weight | 8weeks after intervention
  Body weight assessed by blood test after 2-week use of CGM and dietary education
Pre- and post-intervention questionnaire: Diabetes Treatment Satisfaction Questionnaire (DTSQ) | 8weeks after intervention
  Pre- and post-intervention questionnaires, assessed by self-reported survey. The questionnaire is composed of three parts.
  * total satisfaction (minimum 0, maximum 36, higher scores mean a better outcome.)
  * perceived hyperglycaemia (minimum 0, maximum 6, higher scores mean a worse outcome.)
  * perceived hypoglycaemia (minimum 0, maximum 6, higher scores mean a worse outcome.)
Pre- and post-intervention questionnaire: Summary of Diabetes Self-Care Activities Questionnaire (SDSCAS). | 8weeks after intervention
  Pre- and post-intervention questionnaires, assessed by self-reported survey. The questionnaire is composed of five parts.
  * diet (values: minimum 0, maximum 28, higher scores mean a better outcome.)
  * exercise (minimum 0, maximum 14, higher scores mean a better outcome.)
  * blood sugar check-up (values: minimum 0, maximum 14, higher scores mean a better outcome.)
  * foot care (minimum 0, maximum 14, higher scores mean a better outcome.)
  * smoking (minimum 0, maximum 1, higher scores mean a worse outcome.)

CONTACTS AND LOCATIONS:
Overall Officials: Park, Study Director — cydoctor68@gmail.com
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No